CLINICAL TRIAL: NCT06483841
Title: Parents as Partners: Effectiveness of the Program in a Portuguese Sample of Couples During the Transition to Parenthood
Brief Title: Parents as Partners: Effectiveness of the Program in a Portuguese Sample
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade do Porto (Other)
Collaborators: Foundation for Science and Technology, Portugal (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2023/07-17
Record Dates: First submitted 2024-06-17; First posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-05

CONDITIONS: Healthy
Keywords: Randomized clinical trial; Transition to parenthood; Father involvement; Group intervention

STUDY DESIGN:
Intervention Model Description: The Parents as Partners program consists of 8 weekly group sessions attended by couples and was developed to strengthen the coparental relationship and promote paternal involvement. After consenting to their participation, couples will be randomly assigned to one of two conditions: intervention group or waitlist-control group. Participants will be assessed before and after the intervention on (co)parental, dyadic and work-family dimensions. Baseline (before intervention), post-test (2 months after baseline) and a follow-up assessment 6 months after the program will be performed. The intervention group will participate in the program, focusing on 5 family domains: Parents as Individuals; Parent-Child Relationships; Couple Relationship; Family of Origin Patterns; Stressors and Supports. Parents in the waitlist-control group will receive the intervention once their parti
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Testing the Parents as Partners program (Experimental): Couples (n=51) randomly assigned to this arm will go through 8 weekly group sessions of the Parents as Partners program, facilitated by two trained psychologists. Baseline, post-test and follow-up assessments will entail filling questionnaires collecting data on (co)parental, dyadic and work-family dimensions. At post-test, 6-10 couples will participate in an interview to collect information of their perceived usefulness of the intervention.
  Interventions: Behavioral: Parents as Partners
- Wait-list control group (No Intervention): Couples (n=51) randomly assigned to this arm will not have access to the intervention during the 8 weeks period in which the intervention group is participating in the program. and until their participation in the study is finished, i.e., they have completed all assessments. Baseline, post-test and follow-up assessments will entail filling questionnaires collecting data on (co)parental, dyadic and work-family dimensions. After follow-up, this group will be offered to participate in the intervention if they wish to and if positive outcomes are found.

INTERVENTIONS:
Behavioral: Parents as Partners — The Parents as Partners program consists of 8 weekly group sessions attended by couples and was developed to strengthen the coparental relationship and promote paternal involvement. After consenting to their participation, couples will be randomly assigned to one of two conditions: intervention group or waitlist-control group. Participants will be assessed before and after the intervention on (co)parental, dyadic and work-family dimensions. Baseline (before intervention), post-test (2 months after baseline) and a follow-up assessment 6 months after the program will be performed. The intervention group will participate in the program, focusing on 5 family domains: Parents as Individuals; Parent-Child Relationships; Couple Relationship; Family of Origin Patterns; Stressors and Supports. Parents in the waitlist-control group will receive the intervention once their participation in the study is finished and if positive outcomes are found.
  Arms: Testing the Parents as Partners program

SUMMARY:
This study aims to assess the effectiveness of the "Parents as Partners" program (also named "Supporting Father Involvement"; Cowan et al., 2009) in a sample of Portuguese couples going through the transition to parenthood, i.e., with one child up to the age of 3 years old. The program aims to strengthen the coparenting relationship and consists of 2-hour 8 weekly group sessions attended by couples. Using a mixed-method approach, the researchers will conduct a randomized clinical trial aiming to assess the effectiveness of the intervention on primary and secondary outcomes. Lastly, participants' perceptions of the intervention usefulness will be assessed by conducting interviews with couples who participated in the intervention group (Parents as Partners).

DETAILED DESCRIPTION:
This study was approved by the Ethics Committee of the Faculty of Psychology and Education Sciences of the University of Porto (Ref. 023/07-17).

The curriculum and assessment approach of "Parents as Partners" is built on a 5-domain risk and protective model: Parents as Individuals- Their health, mental health and general well-being; Parent-Child Relationships- Fathers' and mothers' age-appropriate parenting strategies; Couple Relationship- How parents manage their conflict and disagreement; coparenting that is more collaborative than undermining; Family of Origin Patterns- Parents' developmental histories with their parents; what is carried over from the past; how to interrupt intergenerational cycles of harsh treatment, abuse, and neglect; Stressors and Supports- Parents' strategies for coping with external stressors and enlisting support from family, friends, the workplace, and social services. The sessions will be led by two psychologists (male and female) who underwent 24-hour training by the Brazelton Touchpoints Center. The program has a 10-dimension fidelity assessment model, which will be complemented by session checklists. Furthermore, the facilitators will participate in weekly monitoring sessions with professionals specialized in the program.

Participants will be recruited from nurseries and private clinics.

After enrolling in the program, group facilitators conduct an initial interview to get to know the couple and clarify any questions they may have about the program. At this moment, couples will be asked to sign a consent form. After consenting to their participation, couples will be randomly assigned to one of two conditions: intervention group or waitlist-control group. The estimated sample size is 51 couples for the waitlist-control and intervention group each (power of .80; α = .05; G*Power 3.1.9.7). Participants will be assessed before and after the intervention on (co)parental, dyadic and work-family interface dimensions. Parents in the waitlist-control group will receive the intervention once their participation in the study is finished and if positive outcomes are found.

Hypotheses Group effects: The intervention group (IG) is expected to show an increase in coparenting relationship quality, parenting efficacy, and a decrease in parental stress compared to the wait-list control group (CG). Additionally, the investigators expect fathers in the IG to show an increase in parental involvement compared to those in the CG. As for secondary outcomes, the IG is expected to show an increase in the quality of the couple relationship, partner responsiveness and family-work enrichment, and a decrease in family-work conflict compared to the CG. Additionally, the researchers expect an improvement in child's social and emotional development.

Actor and partner effects: The improvement in parental indicators (e.g., parenting efficacy, parental stress) is expected to impact one's parental involvement and the partner's perception of partner responsiveness and coparenting relationship quality.

Statistical procedures: Intent to treat analysis will be applied. All data will be included regardless of participation rate. Repeated measures MANCOVA will be used to address within and between effects of the intervention, alongside T-Tests for comparing IG and CG, and controlling for mental health. The Actor-Partner Interdependence Model will be applied to assess actor and partner effects using Hierarchical Linear Modeling.

To assess the perceived usefulness of the intervention, 6-10 couples from the IG will be interviewed together using a semi-structured script after the posttest survey is completed. These interviews will be conducted by a researcher who has not been involved in the implementation of the program.

Participants data will be stored in an encrypted file, saved on a computer, and only accessible to the main researchers of this study. Confidentiality will be guaranteed by attributing an individual code to each participant/couple. Interviews will be recorded and transcribed and transcriptions will be marked with the same code to ensure the association of the collected data.

ELIGIBILITY:
Inclusion Criteria:

* Heterosexual couples
* Both members of a couple accept to participate
* Couples should have only one child who should be up to 3 years of age
* Both members of the couple must have been parents for the first time together, i.e., they cannot have children from previous relationships
* Should live together.

Exclusion Criteria:

* Severe mental health problems,
* Situations of domestic violence,
* Problematic use of alcohol and/or drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-02-20 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Child-Parent Relationship | Change from baseline (pre-test) to follow-up (6 months after the end of the program implementation).
  Child-Parent Relationship Scale - Short Form: Scale ranges from 1 (definitely does not apply) to 5 (definitively applies); Measures two dimensions: Conflict and Closeness
Coparenting Relationship | Change from baseline (pre-test) to follow-up (6 months after the end of the program implementation).
  Coparenting Relationship Scale: Scale ranges from 0 (not true about us) to 6 (very much true about us); Measures seven dimensions: Coparenting agreement, closeness, exposure to conflict, coparenting support, undermining, endorsement of partner parenting and division of labor.

SECONDARY OUTCOMES:
Parental Stress | Change from baseline (pre-test) to follow-up (6 months after the end of the program implementation).
  Parental Stress Scale: Scale ranges from 1 (totally disagree) to 5 (totally agree); Measures four dimensions: Parental rewards, parental stressors, lack of control and parental satisfaction.
Parenting Efficacy | Change from baseline (pre-test) to follow-up (6 months after the end of the program implementation).
  Parenting Sense of Competence Scale: Scale ranges from 1 (strongly disagree) to 6 (strongly agree); Measures two dimensions: satisfaction and parenting effectiveness
Family-Work Conflict | Change from baseline (pre-test) to follow-up (6 months after the end of the program implementation).
  Work-Family Conflict Scale: Scale ranges from 1 (strongly disagree) to 5 (strongly agree)
Family-Work Enrichment | Change from baseline (pre-test) to follow-up (6 months after the end of the program implementation).
  Work-Family Enrichment Scale: Scale ranges from 1 (strongly disagree) to 5 (strongly agree)
Quality of the Couple Relationship | Change from baseline (pre-test) to follow-up (6 months after the end of the program implementation).
  Quality of Marriage Index: Scale ranges from 1 (very strongly disagree) to 7 (very strongly agree)
Partner Responsiveness | Change from baseline (pre-test) to follow-up (6 months after the end of the program implementation).
  Responsiveness Scale: Scale ranges from 1 (strongly disagree) to 7 (strongly agree)
Child's Social and Emotional Development | Change from baseline (pre-test) to follow-up (6 months after the end of the program implementation).
  Brief Infant-Toddler Social and Emotional Assessment: Scale ranges from 1 (nothing like him/her) to 5 (exactly like him/her)

OTHER OUTCOMES:
Perceived usefulness of the program | Post-test (immediately after the program)
  Semi-structured interview with couples who participated in the IG

CONTACTS AND LOCATIONS:
Overall Officials: Carolina Garraio, MsC, Principal Investigator — PhD Candidate
Locations (1):
- Faculty of Psychology and Educational Sciences of the University of Porto, Porto, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] undefined